CLINICAL TRIAL: NCT06218966
Title: Usability of the Intracochlear Catheter INCAT - a Feasibility Study
Acronym: INCAT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INCAT
Record Dates: First submitted 2023-09-06; First posted 2024-01-23 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2023-09

CONDITIONS: Hearing Loss, Sensorineural; Hearing Loss, Cochlear
Keywords: hearing preservation; cochlear implant; intracochlear catheter; steroids; INCAT; sensorineural hearing loss
MeSH Terms: conditions — Hearing Loss, Sensorineural

STUDY DESIGN:
Intervention Model Description: feasibility study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- study group with INCAT (Experimental): study group with patients receiving intracochlear steroid treatment with the intracochlear catheter INCAT prior to application of the cochlear implant electrode array
  Interventions: Device: intracochlear catheter

INTERVENTIONS:
Device: intracochlear catheter — intracochlear administration of steroids through the intracochlear catheter INCAT

SUMMARY:
This is a feasibility study for a inner ear catheter which will be used to apply steroids to the inner ear. It will be used on nearly deaf patients during their surgery, when they receive an implant that will restore the hearing. Treatment with steroids will improve the maintenance of residual hearing, which will be tested during and after the surgery.

DETAILED DESCRIPTION:
Study Device: The INCAT is an intracochlear catheter which is eligible in Canada for intracochlear drug delivery.

Summary: 24 patients with moderate to profound hearing loss and indication for cochlear implantation will receive intracochlear treatment with steroids with an intracochlear catheter (INCAT) for hearing preservation prior to insertion of the cochlear implant array. Subjects will be considered for the study if they are 18 years of age or older and demonstrate a CNC word score in quiet of 60% or less in the ear to be implanted. Subjects will be followed for 6 months post-activation of the audio processor.

Primary Objectives: Determination of feasibility of the intracochlear catheter INCAT and hearing preservation of residual hearing thresholds intra-, postoperatively, and long-term.

Secondary Objectives: Assessment of quality of life, tinnitus and development of speech perception with the implant up to one year after implantation.

Study Endpoint: Feasibility of using the INCAT and assessment of hearing preservation of residual hearing thresholds. Impedance field telemetry will help to assess hearing thresholds pre-, peri-, and postinsertion.

ELIGIBILITY:
Inclusion Criteria:

* Adults, 18 years of age or older at the time of implantation
* Moderate to profound hearing loss in the low frequencies and severe to profound hearing
* Loss in the high frequencies, bilaterally as defined by (see Figure 4A and B below for example audiogram information)

  * Low-frequency pure tone average (PTA - 250, 500, and 1000 Hz) greater than 40 dB
  * High-frequencies not better than 65 decibels (3000 Hz - 8000 Hz)
* Sensorineural hearing loss, demonstrated by an air-bone gap of less than or equal to 10 dB
* Limited benefit from appropriately fit hearing aids, defined by consonant-nucleus-consonant (CNC) word score in quiet of 60% or less in the ear to be implanted and 70% or less in the non-implanted ear
* CNC word score in quiet of greater than or equal to 10% in the ear to be implanted
* Fluent in English
* No radiological contraindications
* Ability to undergo general anesthesia
* Appropriate motivation and expectation levels
* Stated willingness to comply with all study procedures for the duration of the study
* Able to perform subjective hearing tests
* Able to fill out questionnaires

Exclusion Criteria:

* Age less than 18 years
* Not willing to provide informed consent
* Unable to perform subjective hearing tests
* Unable to fill out questionnaires
* Previous unsensitivity to the investigated drug
* Unable to follow the protocol for any reasons
* Evidence that hearing loss is retrocochlear in origin
* Active middle ear infection
* Skin or scalp condition precluding use of external audio processor
* Suspected cognitive impairment or organic brain dysfunction
* History of prior use of a hearing implant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-01-15 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Pure tone average with air and bone conduction | 12 Months
  air and bone conduction of the frequencies 0.25, 0.5, 1, 2, 4, 6, 8 kHz
speech audiometry | 12 months
  CNC, AzBio, HINT
Impedance | 12 months
  Impedance testing for all electrodes
ECAPs | 12 months
  electrically evoked compound action potential testing for all electrodes
ECochG | 12 months
  electrocochleargraphy

SECONDARY OUTCOMES:
Tinnitus | 12 Months
  Assessment of tinnitus with Tinnitus Handicap Inventory, which is a 25-item self-report measure to determine perceived tinnitus handicap severity

CONTACTS AND LOCATIONS:
Locations (1):
- Sunnybrook Health Sciences Centre Otolaryngology Department, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
on request
Supporting Information: Study Protocol, SAP, ICF
Time Frame: in 12 months and for 12 months
Access Criteria: please contact the PI

REFERENCES:
- [Background] Yildiz E, Gadenstaetter AJ, Gerlitz M, Landegger LD, Liepins R, Nieratschker M, Glueckert R, Staecker H, Honeder C, Arnoldner C. Investigation of inner ear drug delivery with a cochlear catheter in piglets as a representative model for human cochlear pharmacokinetics. Front Pharmacol. 2023 Mar 9;14:1062379. doi: 10.3389/fphar.2023.1062379. eCollection 2023. PMID 36969846
- [Background] Prenzler NK, Salcher R, Timm M, Gaertner L, Lenarz T, Warnecke A. Intracochlear administration of steroids with a catheter during human cochlear implantation: a safety and feasibility study. Drug Deliv Transl Res. 2018 Oct;8(5):1191-1199. doi: 10.1007/s13346-018-0539-z. PMID 29761349
- [Background] Prenzler NK, Salcher R, Lenarz T, Gaertner L, Warnecke A. Dose-Dependent Transient Decrease of Impedances by Deep Intracochlear Injection of Triamcinolone With a Cochlear Catheter Prior to Cochlear Implantation-1 Year Data. Front Neurol. 2020 Apr 15;11:258. doi: 10.3389/fneur.2020.00258. eCollection 2020. PMID 32390924